CLINICAL TRIAL: NCT05488938
Title: An Intensive Anti-Scoliosis Postural Intervention Supported by an Application for Individuals With Rett Syndrome
Brief Title: Intensive Anti-Scoliosis Postural Intervention for Individuals With Rett Syndrome Supported by a Smartphone Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: ASST Santi Paolo e Carlo (Other)
Responsible Party: Principal Investigator, Meir Lotan, Professor, Ariel University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AU-HEA-ML-20201019
Record Dates: First submitted 2022-08-01; First posted 2022-08-05 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Rett Syndrome
Keywords: Rett Syndrome; Scoliosis; Exercise Therapy; Physical Therapy Modalities
MeSH Terms: conditions — Rett Syndrome; Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The orthopedic surgeons who will evaluate the participants' Cobb's angle will be blinded concerning the group to which each participant was assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Group 1) (Experimental): Group 1 will start the rehabilitative intervention immediately after the first evaluation (T1) and carry it out for 10 months with remote supervision until the second evaluation meeting (T2). Then they will be invited to continue the intervention for the next 10 months (between T2 and T3) until the third evaluation meeting but without remote supervision.
  Interventions: Other: Rehabilitative Intervention
- Delayed intervention (Group 2) (Experimental): Group 2 will not conduct the rehabilitative intervetion between T1 and T2. They will start the rehabilitative intervention immediately after the second evaluation (T2) and carry it out for 10 months with remote supervision until the third evaluation meeting (T2).
  Interventions: Other: Rehabilitative Intervention

INTERVENTIONS:
Other: Rehabilitative Intervention — Each program will require the daily performance of different postures and therapeutic activities at the girls' educational facilities and homes, based on the availability of families, for 10 months. Specific strategies that will be implemented will include maintaining asymmetrical postures that oppose the scoliosis curve during activities and exercises in sitting, standing, and walking positions (according to each participant's functional abilities). These strategies refer to a hypercorrective postural positioning of scoliosis. In addition, activities involving weight bearing on the lower limbs, such as walking and standing for at least two hours a day, will be encouraged, and passive stretching and spinal mobilization exercises will be conducted.

SUMMARY:
Background: Scoliosis is the most common orthopedic comorbidity in Rett syndrome (RTT), with a prevalence of 94% and a mean curve progression of 14-21° Cobb annually. A scoliosis prevention intervention based on daily activity programs was proposed for people with RTT within uncontrolled study designs.

Aim: The current study aims to evaluate the effectiveness of a home-based activity program carried out during daily life to slow the progression of scoliosis in girls with RTT.

Ethics: The proposal was approved by Ariel university IRB. All participants' parents will sign informed consent forms.

Participants: Twenty Italian girls aged between six and 16 years with a genetically confirmed classic RTT and scoliosis at a severity level between 10° and 40° Cobb will be recruited and randomly divided into two groups (immediate intervention - Group 1; wait-list-intervention - Group 2). Both groups will follow the same 10-month intervention program, 10 months apart.

Outcome measures: Participants' scoliosis Cobb's angle, motor functioning, and behavioral characteristics will be assessed three times.

Procedure: Each participant will be evaluated three times: at T1, T2, and T3. Participants in the Group 1 will conduct the intervention for 10 months between T0 and T1. Group 2 will perform the intervention between T1 and T2. The interventions will comprise daily home-based activity programs carried out by participants' caregivers within everyday living environments. An expert therapist will remotely supervise each program through an ad hoc developed smartphone application. Specific strategies that will be implemented during the intervention will include the maintenance of asymmetrical postures that oppose the scoliosis curve during activities and exercises in sitting, standing, and walking positions (according to each participant's functional abilities). These strategies refer to a hypercorrective postural positioning of scoliosis. In addition, activities involving weight bearing on the lower limbs, such as walking and standing for at least two hours a day, will be encouraged, and passive stretching and spinal mobilization exercises will be conducted.

DETAILED DESCRIPTION:
Study Aims The current study aims to evaluate the effectiveness of an anti-scoliotic physiotherapy program carried out during daily life and focuses on hypercorrective postures and increasing the level of activity to assess whether or not it is possible to slow the progression of scoliosis in girls with Rett syndrome (RTT).

The current research project has the following research objectives:

* Primary objectives:

  1. Build, implement and evaluate a physiotherapy program for contrasting scoliosis trajectory adapted to individuals with RTT;
  2. Develop a secondary deformity prevention program through early intervention for people with RTT.
* Secondary objectives:

  1. Build and evaluate the efficiency of a support application for carrying out rehabilitation exercises;
  2. Explore the factors influencing adherence and implementation of intervention from the perspective of both families and therapists in light abovementioned applicationd above.

Study Design A randomized controlled study with a waiting list design will be applied.

Ethical Issues The Ariel University Institutional Review Board (IRB) approved the study (no. AU-HEA-ML-20201019) that will be conducted according to the ethical principles of the Helsinki Declaration and local regulations. All details relating to the study procedure will be discussed with participants' parents or legal representatives, and an informed consent form will be signed for participation. Enrolment will be voluntary, with participants not receiving any financial or otherwise incentives for participation.

Study Population According to a sample size calculation analysis, a group of 20 girls aged between six and 16 years with genetically confirmed classic RTT and scoliosis will be recruited from the San Paolo Hospital (Milan, Italy) or the Italian Rett Association (AIRett - Verona, Italy).

Procedure The participants' parents will receive an information sheet regarding the study and informed consent for participating and collecting video materials at the recruitment. A reference telephone number and an e-mail address will be provided to be contacted in case they would like further information or would like to communicate the exit from the study. The eligibility of the candidates will be assessed at the time of recruitment (T1) through an initial neurological or physiatrist evaluation. At the same time, each participant will undergo a rehabilitation evaluation to collect the outcome measures (see section "Data collection") and create an individualized intervention plan specific to the participant's scoliosis, functional abilities, and parental/educational setting's availability. During the evaluation, the postural needs of the participants will also be identified, and a qualified technician will build or adjust the positioning devices, making them suitable for each intervention plan. Participating girls will be randomly divided into treatment (Group 1) or delayed treatment (Group 2) groups using block randomization. Participants in Group 1 will begin carrying out the rehabilitation program immediately after the first assessment session (T1). Each program will require the daily performance of different postures and therapeutic activities at the girls' educational facilities and homes, based on the availability of families, for 10 months. Specific strategies that will be implemented will include maintaining asymmetrical postures that oppose the scoliosis curve during activities and exercises in sitting, standing, and walking positions (according to each participant's functional abilities). These strategies refer to a hypercorrective postural positioning of scoliosis. In addition, activities involving weight bearing on the lower limbs, such as walking and standing for at least two hours a day, will be encouraged, and passive stretching and spinal mobilization exercises will be conducted.

Participants' parents and local reference physiotherapists who will supervise the program in the educational or home setting will be involved in training sessions to learn the performance of the child's program activities. In addition, a smartphone "ActivRett" activity application will be constructed for this research. The application will be downloaded and used by the group that takes care of each participant. It will contain the participant's individualized therapeutic indications and allow the collection of data relating to the development and execution of the program. Further support for parents, caregivers, and therapists will be provided via Skype by an Italian therapist (AR) experienced in treating individuals with RTT at the program's start and every two months. These meetings will discuss the program's progress, solve problems, reorganize schedules, adjust the suggested exercises, assess the achievement of objectives, and if needed, set other goals.

At the end of the intervention of Group 1 (10 months after its start), the outcome measures will be collected again for all participants (T2), and those in group 1 will be allowed to continue using the application without receiving the Skype mentioned above calls. Then, those included in Group 2 will be reevaluated and actively participate in the planned intervention, which will be carried out for the second period of 10 months. At the end of the intervention phase of Group 2, the outcome measures will be collected again for all participants (T3), and the data obtained will be analyzed by the researchers. At the end of each intervention phase, a specific questionnaire will be administered to the parents, therapists, teachers, and other caregivers involved in the intervention program mentioned above to assess the participants' satisfaction with different aspects of the intervention.

Data analysis The normality of each variable's distribution will be assessed using the Shapiro-Wilk normality test. The ages, amount of received physical rehabilitation interventions, scoliotic curve degrees, behavioral characteristics, and activity and gross motor functional levels obtained at T1 will be compared between the two groups to assess their comparability through Wilcoxon's signed-rank test or Student's T-test (dependent of the variable distribution characteristics). Changes in the variables of each group at T1, T2, and T3 will be evaluated with Friedman's test or with the repeated measure ANOVA (dependent on the variable distribution characteristics). Between groups comparison for each variable collected at T1, T2, and T3 and for their variations that occurred between T1 and T2 and between T2 and T3 will be conducted using the Wilcoxon's signed-rank test or Student's T-test (dependent on the variable distribution characteristics), applying an appropriate adjustment for the age and gross motor skills of the participants. Relations will be searched between variables collected at T1 and the changes in the scoliosis curve degree and motor functioning after the treatment using Spearman's rank correlation coefficient or Pearson's correlation coefficient (dependent on the variable distribution characteristics). Moreover, a relation between the compliance with the proposed program and the changes in the scoliosis curve degree and motor functioning after the treatment will be searched using Spearman's rank correlation coefficient or Pearson's correlation coefficient (dependent on the variable distribution characteristics). The threshold for significance of the above-described analyses will be set at α = 0.05. No correction for multiple comparisons will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RTT with confirmed MECP2 gene mutation;
* Diagnosis of unstructured flexible scoliosis (Cobb angle between 10° and 40°) measured radiologically with an x-ray performed no more than six months before the recruitment;
* Age between 6 and 16 years.

Exclusion Criteria:

* Presence of psychomotor developmental deficit evidenced in the first six months of life or diseases of neurometabolic, infectious, or secondary brain damage trauma origin;
* Previous surgical intervention to the spine or its planning within the study period;
* Use of a corset during most waking hours;
* Clinical judgment of the evaluating specialist doctor who certifies unstable health conditions that are not compatible with the performance of the rehabilitation program (e.g., ongoing or recurrent infections, severe gastrointestinal disorders, drug-resistant epilepsy with multi-day seizures).
* Clinical judgment of the research team suggesting an inability of the home environment to perform the intervention program (change in residence, a planned pregnancy, a pre-planned complex surgical/medical procedure within the period of the planned intervention program for the child or family member) within the intervention period.

Ages: 6 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Scoliosis progression | Three days 10 months apart from each other, before the start of the Group 1 intervention (T1), before the start of the Group 2 intervention (T2), and at the end of the Group 2 intervention (T3).
  The progression of scoliosis will be assessed for each participant by measuring the differences between Cobb's angle measured on three anteroposterior X-rays of the spine collected before and after the intervention of each group. The Cobb's angle will be obtained from the average value of three measurements carried out by independent blinded (to the treatment status of each subject) medical specialists with clinical experience concerning scoliosis in Rett syndrome.
Adherence to the Program | 10 months during the Group 1 intervention phase.
  Adherence to the Program refers to the amount of treatment conducted by the participants compared to the total amount of treatment established in their program. It will be measured by the ad hoc developed smartphone application which will record the percentage of the performance of each activity foreseen in the programs.
Adherence to the Program | 10 months during the Group 2 intervention phase.
  Adherence to the Program refers to the amount of treatment conducted by the participants compared to the total amount of treatment established in their program. It will be measured by the ad hoc developed smartphone application which will record the percentage of the performance of each activity foreseen in the programs.

SECONDARY OUTCOMES:
Gross Motor Function Level | 30 minutes, before the beginning of the Group 1 intervention.
  The gross motor function level, including the ability to walk, will be measured for each participant during the rehabilitation assessments using the Rett Syndrome Motor Evaluation Scale. This scale includes 25 items that examine motor function divided into six sections: standing, sitting, postural transfers, walking, running, and climbing / descending stairs. Sixteen items are rated on a discrete scale, ranging from 0 (indicates no or very mild impairment) and 4 (severe impairment). Nine items related to walking skills are evaluated on a discrete scale with a score from 0 to 2 where 0 indicates that the activity could always be completed by the subject and 2 that is assigned if the item cannot be carried out. The items' scores are added together, thus giving a total RESMES score (range: 0 to 82). Moreover, a score for each section can be calculated.
Gross Motor Function Level | 30 minutes, before the beginning of the Group 2 intervention.
  The gross motor function level, including the ability to walk, will be measured for each participant during the rehabilitation assessments using the Rett Syndrome Motor Evaluation Scale. This scale includes 25 items that examine motor function divided into six sections: standing, sitting, postural transfers, walking, running, and climbing / descending stairs. Sixteen items are rated on a discrete scale, ranging from 0 (indicates no or very mild impairment) and 4 (severe impairment). Nine items related to walking skills are evaluated on a discrete scale with a score from 0 to 2 where 0 indicates that the activity could always be completed by the subject and 2 that is assigned if the item cannot be carried out. The items' scores are added together, thus giving a total RESMES score (range: 0 to 82). Moreover, a score for each section can be calculated.
Gross Motor Function Level | 30 minutes, at the end of the Group 2 intervention.
  The gross motor function level, including the ability to walk, will be measured for each participant during the rehabilitation assessments using the Rett Syndrome Motor Evaluation Scale. This scale includes 25 items that examine motor function divided into six sections: standing, sitting, postural transfers, walking, running, and climbing / descending stairs. Sixteen items are rated on a discrete scale, ranging from 0 (indicates no or very mild impairment) and 4 (severe impairment). Nine items related to walking skills are evaluated on a discrete scale with a score from 0 to 2 where 0 indicates that the activity could always be completed by the subject and 2 that is assigned if the item cannot be carried out. The items' scores are added together, thus giving a total RESMES score (range: 0 to 82). Moreover, a score for each section can be calculated.
Behavioral Characteristics | 15 minutes, before the beginning of the Group 1 intervention.
  The behavioral characteristics of the participants will be evaluated through the Rett Syndrome Behavior Questionnaire (RSBQ) administration. The RSBQ is a questionnaire created by comparing the behavioral aspects of people with Rett syndrome with those of individuals with severe intellectual disability. The questionnaire is filled in by parents who are asked to provide an evaluation of the behavioral characteristics shown by their child at the time of completion. The RSBQ includes elements describing behavioral characteristics and assessing physical capabilities, including hand function, sitting, and walking skills. Other items evaluated by the questionnaire include sleep disturbances, respiratory difficulties, mood disturbances, self-harm, social skills, and stereotyped hand movements. The RSBQ comprises 45 items scored on a three-point Likert scale (0 - Not true; 2 - Very or often true), providing a total score between 0 and 90 points.
Behavioral Characteristics | 15 minutes, before the beginning of the Group 2 intervention.
  The behavioral characteristics of the participants will be evaluated through the Rett Syndrome Behavior Questionnaire (RSBQ) administration. The RSBQ is a questionnaire created by comparing the behavioral aspects of people with Rett syndrome with those of individuals with severe intellectual disability. The questionnaire is filled in by parents who are asked to provide an evaluation of the behavioral characteristics shown by their child at the time of completion. The RSBQ includes elements describing behavioral characteristics and assessing physical capabilities, including hand function, sitting, and walking skills. Other items evaluated by the questionnaire include sleep disturbances, respiratory difficulties, mood disturbances, self-harm, social skills, and stereotyped hand movements. The RSBQ comprises 45 items scored on a three-point Likert scale (0 - Not true; 2 - Very or often true), providing a total score between 0 and 90 points.
Behavioral Characteristics | 15 minutes, at the end of the Group 2 intervention.
  The behavioral characteristics of the participants will be evaluated through the Rett Syndrome Behavior Questionnaire (RSBQ) administration. The RSBQ is a questionnaire created by comparing the behavioral aspects of people with Rett syndrome with those of individuals with severe intellectual disability. The questionnaire is filled in by parents who are asked to provide an evaluation of the behavioral characteristics shown by their child at the time of completion. The RSBQ includes elements describing behavioral characteristics and assessing physical capabilities, including hand function, sitting, and walking skills. Other items evaluated by the questionnaire include sleep disturbances, respiratory difficulties, mood disturbances, self-harm, social skills, and stereotyped hand movements. The RSBQ comprises 45 items scored on a three-point Likert scale (0 - Not true; 2 - Very or often true), providing a total score between 0 and 90 points.
Caregivers' Burden | 15 minutes, at the end of the Group 1 intervention.
  The burden related to the implementation of the treatment will be assessed through the administration, at the of each intervention phase, of an ad hoc developed questionnaire to all parents, therapists, teachers, and other caregivers involved in the intervention. The items included in this questionnaire will address the burden derived from the treatment implementation, the parental satisfaction, and the intervention's perceived efficacy concerning functional skills and the trunk and spine posture. The questionnaire comprises 10 items scored on a five-point Likert scale (0 - Completely disagree; 4 - Completely agree), providing a total score between 0 and 50 points.
Caregivers' Burden | 15 minutes, at the end of the Group 2 intervention.
  The burden related to the implementation of the treatment will be assessed through the administration, at the of each intervention phase, of an ad hoc developed questionnaire to all parents, therapists, teachers, and other caregivers involved in the intervention. The items included in this questionnaire will address the burden derived from the treatment implementation, the parental satisfaction, and the intervention's perceived efficacy concerning functional skills and the trunk and spine posture. The questionnaire comprises 10 items scored on a five-point Likert scale (0 - Completely disagree; 4 - Completely agree), providing a total score between 0 and 50 points.

CONTACTS AND LOCATIONS:
Overall Officials: Meir Lotan, PhD, Principal Investigator — Department of Physiotherapy, School of Health Sciences, Ariel University
Locations (1):
- Centro AIRETT Ricerca e Innovazione (CARI), Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
The investigators plan to share the anonymized IPD related to participants' age, level of Rett syndrome severity, Scoliosis Progression, Adherence to the Program, Gross Motor Function Level, Behavioral Characteristics, and Caregivers' Burden. The information will be attached to scientific articles published after the study ends as supplementary materials.
Time Frame: The IPD will be available if and when scientific articles related to this study are published. Should the data be published, they will be available indefinitely in the scientific literature.
Access Criteria: The investigators plan to submit scientific articles related to the present study to be published in an open access peer-review scientific journal. Therefore, if the articles are published, the data will be available on the website of the journal in which they were published.

REFERENCES:
- [Background] Amir RE, Van den Veyver IB, Wan M, Tran CQ, Francke U, Zoghbi HY. Rett syndrome is caused by mutations in X-linked MECP2, encoding methyl-CpG-binding protein 2. Nat Genet. 1999 Oct;23(2):185-8. doi: 10.1038/13810. PMID 10508514
- [Background] Fombonne E, Simmons H, Ford T, Meltzer H, Goodman R. Prevalence of pervasive developmental disorders in the British nationwide survey of child mental health. Int Rev Psychiatry. 2003 Feb-May;15(1-2):158-65. doi: 10.1080/0954026021000046119. PMID 12745327
- [Background] Skjeldal OH, von Tetzchner S, Aspelund F, Herder GA, Lofterld B. Rett syndrome: geographic variation in prevalence in Norway. Brain Dev. 1997 Jun;19(4):258-61. doi: 10.1016/s0387-7604(97)00572-x. PMID 9187475
- [Background] Pini G, Milan M, Zappella M. Rett syndrome in northern Tuscany (Italy): family tree studies. Clin Genet. 1996 Dec;50(6):486-90. doi: 10.1111/j.1399-0004.1996.tb02718.x. PMID 9147879
- [Background] Logan SW, Huang HH, Stahlin K, Galloway JC. Modified ride-on car for mobility and socialization: single-case study of an infant with Down syndrome. Pediatr Phys Ther. 2014 Winter;26(4):418-26. doi: 10.1097/PEP.0000000000000070. PMID 25192001
- [Background] Hagberg B, Witt-Engerstrom I. Rett syndrome: a suggested staging system for describing impairment profile with increasing age towards adolescence. Am J Med Genet Suppl. 1986;1:47-59. doi: 10.1002/ajmg.1320250506. PMID 3087203
- [Background] Bassett GS, Tolo VT. The incidence and natural history of scoliosis in Rett syndrome. Dev Med Child Neurol. 1990 Nov;32(11):963-6. doi: 10.1111/j.1469-8749.1990.tb08118.x. PMID 2269405
- [Background] Ager S, Downs J, Fyfe S, Leonard H. Parental experiences of scoliosis management in Rett syndrome. Disabil Rehabil. 2009;31(23):1917-24. doi: 10.1080/09638280902846392. PMID 19479541
- [Background] Ager S, Fyfe S, Christodoulou J, Jacoby P, Schmitt L, Leonard H. Predictors of scoliosis in Rett syndrome. J Child Neurol. 2006 Sep;21(9):809-13. doi: 10.1177/08830738060210091501. PMID 16970893
- [Background] Riise R, Brox JI, Sorensen R, Skjeldal OH. Spinal deformity and disability in patients with Rett syndrome. Dev Med Child Neurol. 2011 Jul;53(7):653-7. doi: 10.1111/j.1469-8749.2011.03935.x. Epub 2011 Apr 18. PMID 21501153
- [Background] Lidstrom J, Stokland E, Hagberg B. Scoliosis in Rett syndrome. Clinical and biological aspects. Spine (Phila Pa 1976). 1994 Jul 15;19(14):1632-5. doi: 10.1097/00007632-199407001-00013. PMID 7940001
- [Background] Downs J, Bergman A, Carter P, Anderson A, Palmer GM, Roye D, van Bosse H, Bebbington A, Larsson EL, Smith BG, Baikie G, Fyfe S, Leonard H. Guidelines for management of scoliosis in Rett syndrome patients based on expert consensus and clinical evidence. Spine (Phila Pa 1976). 2009 Aug 1;34(17):E607-17. doi: 10.1097/BRS.0b013e3181a95ca4. PMID 19644320
- [Background] Percy AK, Lee HS, Neul JL, Lane JB, Skinner SA, Geerts SP, Annese F, Graham J, McNair L, Motil KJ, Barrish JO, Glaze DG. Profiling scoliosis in Rett syndrome. Pediatr Res. 2010 Apr;67(4):435-9. doi: 10.1203/PDR.0b013e3181d0187f. PMID 20032810
- [Background] Huang TJ, Lubicky JP, Hammerberg KW. Scoliosis in Rett syndrome. Orthop Rev. 1994 Dec;23(12):931-7. PMID 7885724
- [Background] Killian JT, Lane JB, Lee HS, Skinner SA, Kaufmann WE, Glaze DG, Neul JL, Percy AK. Scoliosis in Rett Syndrome: Progression, Comorbidities, and Predictors. Pediatr Neurol. 2017 May;70:20-25. doi: 10.1016/j.pediatrneurol.2017.01.032. Epub 2017 Feb 7. PMID 28347601
- [Background] Harrison DJ, Webb PJ. Scoliosis in the Rett syndrome: natural history and treatment. Brain Dev. 1990;12(1):154-6. doi: 10.1016/s0387-7604(12)80200-2. PMID 2344012
- [Background] Downs J, Torode I, Wong K, Ellaway C, Elliott EJ, Christodoulou J, Jacoby P, Thomson MR, Izatt MT, Askin GN, McPhee BI, Bridge C, Cundy P, Leonard H. The Natural History of Scoliosis in Females With Rett Syndrome. Spine (Phila Pa 1976). 2016 May;41(10):856-63. doi: 10.1097/BRS.0000000000001399. PMID 26679887
- [Background] Neul JL, Fang P, Barrish J, Lane J, Caeg EB, Smith EO, Zoghbi H, Percy A, Glaze DG. Specific mutations in methyl-CpG-binding protein 2 confer different severity in Rett syndrome. Neurology. 2008 Apr 15;70(16):1313-21. doi: 10.1212/01.wnl.0000291011.54508.aa. Epub 2008 Mar 12. PMID 18337588
- [Background] Mehta J, Gibson M. The treatment of neuromuscular scoliosis. Current Orthopaedics. 2003; 17(4): 313-21. doi:10.1016/S0268-0890(03)00002-1.
- [Background] Westerlund LE, Gill SS, Jarosz TS, Abel MF, Blanco JS. Posterior-only unit rod instrumentation and fusion for neuromuscular scoliosis. Spine (Phila Pa 1976). 2001 Sep 15;26(18):1984-9. doi: 10.1097/00007632-200109150-00008. PMID 11547196
- [Background] Rocos B, Zeller R. Correcting Scoliosis in Rett Syndrome. Cureus. 2021 Jun 3;13(6):e15411. doi: 10.7759/cureus.15411. eCollection 2021 Jun. PMID 34249558
- [Background] Barney CC, Merbler AM, Quest K, Byiers BJ, Wilcox GL, Schwantes S, Roiko SA, Feyma T, Beisang A, Symons FJ. A case-controlled comparison of postoperative analgesic dosing between girls with Rett syndrome and girls with and without developmental disability undergoing spinal fusion surgery. Paediatr Anaesth. 2017 Mar;27(3):290-299. doi: 10.1111/pan.13066. Epub 2017 Feb 8. PMID 28177174
- [Background] Larsson EL, Aaro S, Ahlinder P, Normelli H, Tropp H, Oberg B. Long-term follow-up of functioning after spinal surgery in patients with Rett syndrome. Eur Spine J. 2009 Apr;18(4):506-11. doi: 10.1007/s00586-008-0876-6. Epub 2009 Jan 23. PMID 19165511
- [Background] Downs J, Young D, de Klerk N, Bebbington A, Baikie G, Leonard H. Impact of scoliosis surgery on activities of daily living in females with Rett syndrome. J Pediatr Orthop. 2009 Jun;29(4):369-74. doi: 10.1097/BPO.0b013e3181a53b41. PMID 19461379
- [Background] Downs J, Torode I, Wong K, Ellaway C, Elliott EJ, Izatt MT, Askin GN, Mcphee BI, Cundy P, Leonard H; Rett syndrome spinal fusion group. Surgical fusion of early onset severe scoliosis increases survival in Rett syndrome: a cohort study. Dev Med Child Neurol. 2016 Jun;58(6):632-8. doi: 10.1111/dmcn.12984. Epub 2015 Dec 11. PMID 26661519
- [Background] Kerr AM, Webb P, Prescott RJ, Milne Y. Results of surgery for scoliosis in Rett syndrome. J Child Neurol. 2003 Oct;18(10):703-8. doi: 10.1177/08830738030180101201. PMID 14649553
- [Background] Roberts SB, Tsirikos AI. Factors influencing the evaluation and management of neuromuscular scoliosis: A review of the literature. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):613-623. doi: 10.3233/BMR-160675. PMID 26966821
- [Background] SOSORT guideline committee; Weiss HR, Negrini S, Rigo M, Kotwicki T, Hawes MC, Grivas TB, Maruyama T, Landauer F. Indications for conservative management of scoliosis (guidelines). Scoliosis. 2006 May 8;1:5. doi: 10.1186/1748-7161-1-5. PMID 16759357
- [Background] Kotwicki T, Jozwiak M. Conservative management of neuromuscular scoliosis: personal experience and review of literature. Disabil Rehabil. 2008;30(10):792-8. doi: 10.1080/09638280801889584. PMID 18432437
- [Background] Karimi MT, Rabczuk T. Scoliosis conservative treatment: A review of literature. J Craniovertebr Junction Spine. 2018 Jan-Mar;9(1):3-8. doi: 10.4103/jcvjs.JCVJS_39_17. PMID 29755230
- [Background] Haleem S, Nnadi C. Scoliosis: a review. Paediatr Child Health (Oxford) 2018; 28(5): 209-17. doi:10.1016/j.paed.2018.03.007.
- [Background] Ferrari A, Ferrara C, Balugani M, Sassi S. Severe scoliosis in neurodevelopmental disabilities: clinical signs and therapeutic proposals. Eur J Phys Rehabil Med. 2010 Dec;46(4):563-80. PMID 21224789
- [Background] Downs J, Torode I, Ellaway C, Jacoby P, Bunting C, Wong K, Christodoulou J, Leonard H. Family satisfaction following spinal fusion in Rett syndrome. Dev Neurorehabil. 2016;19(1):31-7. doi: 10.3109/17518423.2014.898107. Epub 2014 Apr 11. PMID 24724550
- [Background] Olafsson Y, Saraste H, Al-Dabbagh Z. Brace treatment in neuromuscular spine deformity. J Pediatr Orthop. 1999 May-Jun;19(3):376-9. PMID 10344323
- [Background] Lotan M, Merrick J, Carmeli E. Managing scoliosis in a young child with Rett syndrome: a case study. ScientificWorldJournal. 2005 Mar 29;5:264-73. doi: 10.1100/tsw.2005.33. PMID 15798886
- [Background] Romano A, Ippolito E, Risoli C, Malerba E, Favetta M, Sancesario A, Lotan M, Moran DS. Intensive Postural and Motor Activity Program Reduces Scoliosis Progression in People with Rett Syndrome. J Clin Med. 2022 Jan 22;11(3):559. doi: 10.3390/jcm11030559. PMID 35160011
- [Background] Lotan M, Downs J, Elefant C. A Pilot Study Delivering Physiotherapy Support for Rett Syndrome Using a Telehealth Framework Suitable for COVID-19 Lockdown. Dev Neurorehabil. 2021 Aug;24(6):429-434. doi: 10.1080/17518423.2021.1914762. Epub 2021 Apr 15. PMID 33853477
- [Background] Romano A, Di Rosa G, Tisano A, Fabio RA, Lotan M. Effects of a remotely supervised motor rehabilitation program for individuals with Rett syndrome at home. Disabil Rehabil. 2022 Oct;44(20):5898-5908. doi: 10.1080/09638288.2021.1949398. Epub 2021 Jul 20. PMID 34282992
- [Background] Neul JL, Kaufmann WE, Glaze DG, Christodoulou J, Clarke AJ, Bahi-Buisson N, Leonard H, Bailey ME, Schanen NC, Zappella M, Renieri A, Huppke P, Percy AK; RettSearch Consortium. Rett syndrome: revised diagnostic criteria and nomenclature. Ann Neurol. 2010 Dec;68(6):944-50. doi: 10.1002/ana.22124. PMID 21154482
- [Background] Fabio RA, Martinazzoli C, Antonietti A. Development and standardization of the "RARS"(Rett Assessment Rating Scale). Life Span Disabil 2005; 8(2): 257-81.
- [Background] Romano A, Capri T, Semino M, Bizzego I, Di Rosa G, Fabio RA. Gross Motor, Physical Activity and Musculoskeletal Disorder Evaluation Tools for Rett Syndrome: A Systematic Review. Dev Neurorehabil. 2020 Nov;23(8):485-501. doi: 10.1080/17518423.2019.1680761. Epub 2019 Oct 31. PMID 31668104
- [Background] Rodocanachi Roidi ML, Isaias IU, Cozzi F, Grange F, Scotti FM, Gestra VF, Gandini A, Ripamonti E. Motor function in Rett syndrome: comparing clinical and parental assessments. Dev Med Child Neurol. 2019 Aug;61(8):957-963. doi: 10.1111/dmcn.14109. Epub 2018 Nov 26. PMID 30474854
- [Background] Rodocanachi Roidi ML, Isaias IU, Cozzi F, Grange F, Scotti FM, Gestra VF, Gandini A, Ripamonti E. A New Scale to Evaluate Motor Function in Rett Syndrome: Validation and Psychometric Properties. Pediatr Neurol. 2019 Nov;100:80-86. doi: 10.1016/j.pediatrneurol.2019.03.005. Epub 2019 Mar 16. PMID 31047758
- [Background] Mount RH, Charman T, Hastings RP, Reilly S, Cass H. The Rett Syndrome Behaviour Questionnaire (RSBQ): refining the behavioural phenotype of Rett syndrome. J Child Psychol Psychiatry. 2002 Nov;43(8):1099-110. doi: 10.1111/1469-7610.00236. PMID 12455930
- [Background] Lotan M, Ippolito E, Favetta M, Romano A. Skype Supervised, Individualized, Home-Based Rehabilitation Programs for Individuals With Rett Syndrome and Their Families - Parental Satisfaction and Point of View. Front Psychol. 2021 Sep 16;12:720927. doi: 10.3389/fpsyg.2021.720927. eCollection 2021. PMID 34603144
- [Background] Armstrong RA. When to use the Bonferroni correction. Ophthalmic Physiol Opt. 2014 Sep;34(5):502-8. doi: 10.1111/opo.12131. Epub 2014 Apr 2. PMID 24697967

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT05488938/Prot_SAP_ICF_000.pdf